CLINICAL TRIAL: NCT01290965
Title: A Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics, and Effect of Treatment With SCY 635 on Plasma HCV RNA Following 15 Days of Oral Administration in Adult Patients With Chronic Hepatitis C Infection
Brief Title: Safety, PK and Efficacy of 15 Days of SCY-635 Treatment in Hepatitis C Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCY-635-104
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — SCY-635

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo comparator (Placebo Comparator)
  Interventions: Drug: Placebo
- SCY-635 30 mg once daily (Active Comparator)
  Interventions: Drug: SCY-635
- SCY-635 100 mg once daily (Active Comparator)
  Interventions: Drug: SCY-635
- SCY-635 300 mg once daily (Active Comparator)
  Interventions: Drug: SCY-635
- SCY-635 100 mg three times daily (Active Comparator)
  Interventions: Drug: SCY-635
- SCY-635 200 mg three times daily (Active Comparator)
  Interventions: Drug: SCY-635
- SCY-635 300 mg three times daily (Active Comparator)
  Interventions: Drug: SCY-635

INTERVENTIONS:
Drug: Placebo — Oral tablet given once or three times daily for 15 consecutive days
  Arms: Placebo comparator
Drug: SCY-635 — oral capsule
  Arms: SCY-635 100 mg once daily; SCY-635 100 mg three times daily; SCY-635 200 mg three times daily; SCY-635 30 mg once daily; SCY-635 300 mg once daily; SCY-635 300 mg three times daily

SUMMARY:
This study will examine the effectiveness of 15 days of therapy with SCY-635 in reducing hepatitis C virus (HCV) RNA levels.

ELIGIBILITY:
Inclusion Criteria:

A potential subject will be eligible for participation in this study if he or she meets all of the following inclusion criteria:

* The subject is either male or female, between the ages of 18 and 65 years (inclusive).
* The subject has read and signed a Subject Informed Consent form to participate in the study. If the subject is not fluent in English, the Subject Informed Consent form must be translated into his or her native language.
* Female subjects of childbearing potential (i.e., women not surgically sterile or at least two years postmenopausal) must agree to utilize one of the following forms of contraception from Screening through completion of the study: abstinence, barrier (condom, diaphragm with spermicide), intrauterine device (IUD), or vasectomized partner (six months minimum). Hormonal contraception (oral, transdermal, implant, or injection) is not permitted during the study period (i.e., from Screening through the Follow-up visit). Note: For women aged <50 years, postmenopausal is defined as at least two years cessation of menses. For women aged ≥50 years, postmenopausal is defined as at least one year cessation of menses. Estrogen replacement is allowed during the study.
* The subject exhibits quantifiable plasma levels of HCV-specific RNA in excess of 100,000 IU/mL as determined by the quantitative Roche COBAS taqMan assay.
* The subject has a negative urine screen for amphetamines, barbiturates, cocaine, opiates, and phencyclidine at Screening.
* If female, the subject has a negative serum pregnancy test at Screening (within 30 days prior to dosing) and a negative urine pregnancy test on Study Day -1.

Exclusion Criteria:

A potential subject will be excluded from participation in the study if he or she meets any of the following exclusion criteria:

* The subject has a history of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition which, in the opinion of the Principal Investigator, may jeopardize the safety of the subject or may impact the validity of the study results.
* The subject is infected with any HCV genotype other than genotype 1.
* The subject has documented positive antibody tests for Human Immunodeficiency Virus Types 1 or 2 (p24 antibody specific for HIV-1 or HIV-2) or Hepatitis B virus (HBV) surface antigen (HbSAg) or at Screening exhibits serologic evidence of infection with either HIV-1, HIV-2 or HBV.
* The subject has donated blood within 30 days prior to dosing or donated plasma within 14 days prior to dosing.
* The subject has used any investigational agent within three months prior to dosing.
* The subject has received any FDA-approved anti-HCV therapy (including ribavirin or any product that contains interferon) within three months prior to dosing.
* The subject exhibits evidence of decompensated liver disease, as marked by bilirubin greater than 4 mg/dL, albumin less than 3.0 g/dL, prothrombin time greater than 2 seconds prolonged, or history of bleeding esophageal varices, ascites or hepatic encephalopathy.
* The subject is an organ transplant recipient.
* The subject exhibits ALT values greater than or equal to 2.5 times the upper limit of normal.
* The subject exhibits evidence of hepatocellular carcinoma either by exhibiting a serum alpha-fetoprotein concentration which exceeds 50 mg/L or by exhibiting a mass suggestive of liver cancer by ultrasound or other imaging technology.
* The subject exhibits evidence of ongoing alcohol or substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Plasma HCV RNA level | 22 days
Incidence and severity of treatment-emergent adverse events and changes in laboratory values as measures of safety and tolerability. | 22 days

SECONDARY OUTCOMES:
Pharmacokinetic assessment of SCY-635 | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Heuman, MD, Principal Investigator — McGuire Veterans Affairs Medical Center, Richmond, Virginia; Jacob Lalezari, MD, Principal Investigator — Quest Clinical Research, San Francisco, California
Locations (2):
- United States (2):
  - Quest Clinical Research, San Francisco, California
  - McGuire Veterans Affairs Medical Center, Richmond, Virginia

REFERENCES:
- [Derived] Hopkins S, DiMassimo B, Rusnak P, Heuman D, Lalezari J, Sluder A, Scorneaux B, Mosier S, Kowalczyk P, Ribeill Y, Baugh J, Gallay P. The cyclophilin inhibitor SCY-635 suppresses viral replication and induces endogenous interferons in patients with chronic HCV genotype 1 infection. J Hepatol. 2012 Jul;57(1):47-54. doi: 10.1016/j.jhep.2012.02.024. Epub 2012 Mar 13. PMID 22425702